CLINICAL TRIAL: NCT06726278
Title: Significance of Misoprostol-induced Cervical Ripening Prior to Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hayat Abad Medical Complex, Peshawar (Other Government)
Collaborators: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Madiha Iqbal, Assistant Professor, Hayat Abad Medical Complex, Peshawar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: HMCKP1
Record Dates: First submitted 2024-11-30; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Hysteroscopy; Cervical Ripening
Keywords: Misoprostol; Cervical Ripening; Hysteroscopy; Cervical Dilation
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Although this study is an observational study, masking was used to minimize bias in the assessment of outcomes. The participants were blinded to the group allocation (misoprostol or placebo). Additionally, the care providers performing the hysteroscopic procedures were also blinded to the group assignments to avoid any bias in procedural conduct or outcome reporting.
  The investigators and outcomes assessors involved in the data analysis were also unaware of the group allocation, ensuring impartial evaluation of the results. This blinding process was maintained throughout the study to minimize bias and enhance the reliability of the observed outcomes.
  Since this study does not involve random assignment or an investigational treatment, it is important to note that masking was implemented as part of the observational design to preserve the validity of the findings, despite the lack of intervention assignment typically seen in clinical trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Participants in this group will receive Misoprostol 400 µg, administered orally. This arm is designed to evaluate the efficacy and safety of Misoprostol for the intended clinical outcome.
  Interventions: Drug: Misoprostol 400mcg Tab
- Group B (Placebo Comparator): Participants in this group will receive a placebo that matches the Misoprostol formulation in appearance, but contains no active ingredients. This arm serves as a control to compare the effects of Misoprostol with a non-active substance.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol 400mcg Tab — Misoprostol 400 µg is a synthetic prostaglandin E1 analog used in this clinical trial to evaluate its effects in inducing uterine contractions or labor. This dosage form is typically administered orally, and its primary mechanism involves the softening and dilation of the cervix, making it a common choice in obstetric practices for labor induction. The study will evaluate its efficacy and safety profile when compared to the placebo group. Misoprostol is administered in a single dose of 400 µg, and participants will be monitored for any adverse reactions or labor-related outcomes.
  Arms: Group A
Drug: Placebo — participants will receive a placebo treatment, consisting of an inert substance that has no active pharmacological effect. The placebo is administered in the same manner (vaginally) and at the same time point as Misoprostol, but without any therapeutic action. This group is used to control for potential psychological effects of the intervention, ensuring that any observed
  Arms: Group B

SUMMARY:
The goal of this prospective study is to evaluate the efficacy and safety of misoprostol for cervical ripening prior to hysteroscopy

DETAILED DESCRIPTION:
This prospective study was conducted at Gynecology Department of Hayatabad Medical Complex Peshawar from Aug 2022 to July 2024. Total 539 women's whose elective hysteroscopy was planned were enrolled. Eligible subjects were non-pregnant women between the ages of 18-45, and were confirmed to be so with a negative urine pregnancy test. Before undergoing hysteroscopy, the participants required to have indicators for hysteroscopy (atypical bleeding per vagina and/or infertility; at suspected pathology in utero), with no previous history of surgery or significant cervical pathologies. Exclusion criteria were: any contraindication, such as allergy to prostaglandins, active pelvic infection; severe cardiovascular, hepatic and/or renal disease or previous uterine perforation/cervical incompetence. Approval from Institutional Review Board was obtained under ref # 860. Patients were divided into two groups based on the administration of misoprostol: Group A (n=300) received 400 µg of misoprostol, administered vaginally, 12 hours prior to the scheduled hysteroscopy. Group B (n=239) did not receive misoprostol and served as the control group. Patients and the clinicians who undertook hysteroscopy were blinded to group assignments. It ordered the misoprostol and placebo tablets separately from a hospital pharmacy so they would look identical.

Hysteroscopic Procedure All hysteroscopic procedures were done in the standard conditions with 5.50 mm rigid Hysteroscope (Karl Storz, Germany). The patients were placed in the lithotomy position, and a tenaculum was used to apply anteflexion of the cervix before insertion. The cervical dilation achieved was measured using Hegar dilators in increments of 1 mm until the hysteroscope could be inserted without resistance.

The primary outcome was the amount of cervical dilation achieved on entry to hysteroscopy. The secondary outcomes were: requirement for mechanical dilation, procedure time (from hysteroscope insertion to withdrawal), patient-reported pain score using Visual Analog Scale (VAS) during the procedures, incident of cervical laceration and adverse events including cramping, bleeding per vagina abnormal gastrointestinal discomfort and fever.

Data Collection / analysis Age, parity, and the reason for hysteroscopy were among the baseline demographic data that were gathered. Information was documented during the hysteroscopic procedure, including cervical dilatation, procedure duration, and any complications. Following the surgery, patients used the Visual Analog Scale (VAS) to rate their level of pain. After the surgery, adverse effects were tracked and recorded for up to 24 hours. Using SPSS version 25.0, statistical analysis was carried out, with a significance level set at p-value ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women aged 18-45 years.
* Confirmed non-pregnancy with a negative urine pregnancy test.
* No history of prior surgery or significant cervical pathologies.
* Atypical bleeding per vagina.
* Infertility.
* Suspected uterine pathology.

Exclusion Criteria:

* Contraindications to prostaglandins, such as:
* Allergy to prostaglandins.
* Active pelvic infection.
* Severe cardiovascular, hepatic, and/or renal disease.
* Previous uterine perforation.
* Cervical incompetence.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 539 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Cervical Ripening Success Rate | During the hysteroscopy procedure (up to 30 minutes).
  Proportion of patients achieving adequate cervical dilation with misoprostol alone, defined as a minimum dilation of [specific measure, e.g., 6mm without mechanical dilation].

SECONDARY OUTCOMES:
Requirement for Mechanical Dilation | During the hysteroscopy procedure (up to 30 minutes).
  The proportion of patients requiring additional mechanical dilation during the hysteroscopy procedure.
Procedure Time | During the hysteroscopy procedure (up to 30 minutes).
  Time taken for the entire hysteroscopy procedure, from insertion to withdrawal of the hysteroscope.
VAS Pain Score | Immediately after the hysteroscopy procedure.
  Patient-reported pain scores during the hysteroscopy procedure, assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain).
Incidence of Cervical Lacerations | During the hysteroscopy procedure (up to 30 minutes).
  Proportion of patients experiencing cervical lacerations during the hysteroscopy procedure.
Incidence of Adverse Events | Up to 24 hours after the hysteroscopy procedure.
  Incidence of adverse events, including cramping, bleeding, gastrointestinal discomfort, and fever.

CONTACTS AND LOCATIONS:
Locations (1):
- Hayatabad Medical Complex, Peshawar, Khyber Pukhtoonkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
At this time, individual participant data (IPD) will not be shared due to privacy and confidentiality considerations. The study is focused on internal analysis and reporting of outcomes based on aggregate data. No explicit plan for sharing IPD with other researchers is currently in place, as the focus is on publication of summarized results for public health and clinical advancement